CLINICAL TRIAL: NCT07137364
Title: Efficacy of Spironolactone Combined With Antihypertensive Drugs in Patients With Primary Aldosteronism
Status: Recruiting | Type: Observational
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, Director of the department of Hypertension & Endocrinology, Daping Hospital, Third Military Medical University
Other Study IDs: SPIRO in PA
Record Dates: First submitted 2025-08-03; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Primary Aldosteronism; Hypertension
MeSH Terms: conditions — Hyperaldosteronism; Hypertension | interventions — Spironolactone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unilateral primary aldosteronism group: The patients are diagnosed with unilateral primary aldosteronism based on adrenal venous sampling diagnosis, they will treated with spironolactone according to their own condition
  Interventions: Drug: spironolactone

INTERVENTIONS:
Drug: spironolactone — The patients receive spironolactone treatment based on their conditions
  Other Names: Aldactone

SUMMARY:
The goal of this observational study is to learn about the optimal dose of spironolactone treatment and the long-term outcomes on cardiovascular and cerebrovascular events in patients with lateralized PA who are unwilling to undergo surgery. The main question it aims to answer is:

1. What is the long-term effect of spironolactone treatment for lateralized PA?
2. What is the optimal dose of spironolactone treatment for the relief of renin inhibition in patients with lateralized PA? Participants will receive spironolactone treatment as part of their regular medical care for more than 12 months, and their clinical indicators, including blood pressure, biochemical remission, cardiovascular and renal damage, and the incidence of cardiovascular and cerebrovascular events, will be analyzed.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) is one of the most common causes of endocrine and treatment-resistant hypertension. Current guidelines suggest that surgery and aldosterone receptor antagonists (MRAs), such as spironolactone, are the main treatment for PA. Patients with aldosterone-producing adenoma who decline surgery, as well as those with idiopathic hyperaldosteronism, are usually treated with spironolactone. However, there is a lack of large-scale, long-term, prospective, randomized controlled trials on spironolactone. In a retrospective cohort of 602 PA patients treated with long-term spironolactone therapy, Hundemer et al. found that the 10-year risk of major cardiovascular events and all-cause mortality was increased, compared with that in patients with essential hypertension. In contrast, PA patients who underwent adrenalectomy had a lower risk of cardiorenal vascular events than that in the spironolactone-treated patients, which was comparable to that of patients with essential hypertension. Further analysis revealed that if PA patients remained in a low-renin state after drug therapy, their risk of myocardial infarction, stroke, and heart-failure hospitalization was almost three-fold higher than that in patients with essential hypertension. Therefore, high doses of spironolactone (60~100 mg/d) were recommended to relieve renin suppression. However, prolonged high-dose spironolactone is associated with numerous side effects, including hyperkalaemia, gynaecomastia and sexual dysfunction in men, menstrual irregularities in women, and central-nervous-system symptoms. Moreover, MRAs only block the effect of aldosterone at the receptor level, failing to suppress aldosterone synthesis. In addition, aldosterone exhibits receptor-independent actions. Consequently, whether spironolactone mitigates aldosterone-mediated cardiovascular and cerebrovascular events remains uncertain, and the optimal dose with fewer adverse effects needs to be defined. To clarify the optimal dose of spironolactone treatment and the long-term outcomes on cardiovascular and cerebrovascular events, the researchers conducted a long-term study involving patients with lateralized PA who are unwilling to undergo surgery. When the blood pressure fails to meet the criteria, antihypertensive drugs such as amlodipine and irbesartan, are combined. the PA patients will be confirmed as unilateral PA based on the results of adrenal venous sampling and different doses of spironolactone. The PA patients will take spironolactone treatment as part of their regular medical care for more than 12 months. The blood pressures, biochemical remission, cardiovascular and renal damage, and cardiovascular and cerebrovascular events will be analyzed after the spironolactone treatment. The antihypertensive efficacy and adverse reactions will be studied.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 30~65 years.
2. PA patients with positive screening tests and saline suppression tests, and with AVS to determine lateralization. These patients have hypertension defined as office blood pressure ≥ 140/90 mmHg, or 24-hour ambulatory blood pressure showing average ≥ 130/80 mmHg, daytime blood pressure ≥ 135/85 mmHg, or nighttime blood pressure ≥ 120/70 mmHg.
3. Patients with unilateral aldosterone-producing adenoma who decline surgery, or patients with non-adenoma, unilateral PA confirmed by AVS and meeting the above PA-related hypertension criteria.
4. Provision of written informed consent to participate in the study.

Exclusion Criteria:

1. Hyperkalemia.
2. Renal impairment or have history of renal disease: serum creatinine > 1.5 × upper limit of normal (ULN), dialysis, or nephrotic syndrome.
3. Other confirmed secondary hypertension: pheochromocytoma, Cushing's syndrome, thyroid disorders, parathyroid disorders, acromegaly, renovascular disease, aortic disorders, chronic alcoholism, or drug dependence, etc.
4. Adrenal insufficiency.
5. Heart failure with NYHA class II-IV or stroke.
6. Acute infection, malignancy, severe arrhythmia, psychiatric disorders, or drug/alcohol abuse.
7. Significant hepatic dysfunction or have history of liver disease: AST or ALT > 2 × ULN, cirrhosis, hepatic encephalopathy, esophageal varices or portosystemic shunt.
8. Pregnancy or lactation.
9. Participation in another clinical trial within the past 3 months.
10. Inability to complete follow-up.
11. Refusal to provide informed consent.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change of systolic blood pressure | From enrollment to spironolactone treatment at 12 months.
  This study will gain insight into the effect of spironolactone treatment on systolic blood pressure. The systolic blood pressure (mmHg) is measured before and after spironolactone treatment, respectively. The changes of systolic blood pressure are analyzed after the spironolactone treatment.
Change of diastolic blood pressure | From enrollment to spironolactone treatment at 12 months.
  This study will gain insight into the effect of spironolactone treatment on diastolic blood pressure. The diastolic blood pressure (mmHg) is measured before and after spironolactone treatment, respectively. The changes of diastolic blood pressure are analyzed after the spironolactone treatment.

SECONDARY OUTCOMES:
Change of anti-hypertensive regimen | From enrollment to spironolactone treatment at 12 months.
  This study will gain insight into the effect of spironolactone treatment on anti-hypertensive regimen. The anti-hypertensive regimens are measured before and after spironolactone treatment, respectively. The changes of anti-hypertensive regimens are analyzed after the spironolactone treatment.
Change of serum potassium | From enrollment to spironolactone treatment at 12 months.
  This study will gain insight into the effect of spironolactone treatment on serum potassium. The concentrations of serum potassium (mmol/L) are measured before and after spironolactone treatment, respectively. The changes of serum potassium are analyzed after the spironolactone treatment.
Change of plasma aldosterone | From enrollment to spironolactone treatment at 12 months.
  This study will gain insight into the effect of spironolactone treatment on plasma aldosterone. The concentrations of plasma aldosterone (ng/dL) are measured before and after spironolactone treatment, respectively. The changes of plasma aldosterone are analyzed after the spironolactone treatment.
Change of plasma renin | From enrollment to spironolactone treatment at 12 months.
  This study will gain insight into the effect of spironolactone treatment on plasma renin. The concentrations of plasma renin (mU/L) are measured before and after spironolactone treatment, respectively. The changes of plasma renin are analyzed after the spironolactone treatment.
Change of fasting plasma glucose | From enrollment to spironolactone treatment at 12 months.
  This study will gain insight into the effect of spironolactone treatment on fasting plasma glucose. The concentrations of fasting plasma glucose (mmol/L) are measured before and after spironolactone treatment, respectively. The changes of fasting plasma glucose are analyzed after the spironolactone treatment.
Changes of serum total cholesterol | From enrollment to spironolactone treatment at 12 months.
  This study will gain insight into the effect of spironolactone treatment on serum total cholesterol. The concentrations of serum total cholesterol (mmol/L) are measured before and after spironolactone treatment, respectively. The changes of serum total cholesterol are analyzed after the spironolactone treatment.
Changes of serum triglyceride | From enrollment to spironolactone treatment at 12 months.
  This study will gain insight into the effect of spironolactone treatment on serum triglyceride. The concentrations of serum triglyceride (mmol/L) are measured before and after spironolactone treatment, respectively. The changes of serum triglyceride are analyzed after the spironolactone treatment.
Changes of serum high-density lipoprotein cholesterol | From enrollment to spironolactone treatment at 12 months.
  This study will gain insight into the effect of spironolactone treatment on serum high-density lipoprotein cholesterol. The concentrations of serum high-density lipoprotein cholesterol (mmol/L) are measured before and after spironolactone treatment, respectively. The changes of serum high-density lipoprotein cholesterol are analyzed after the spironolactone treatment.
Changes of serum low-density lipoprotein cholesterol | From enrollment to spironolactone treatment at 12 months.
  This study will gain insight into the effect of spironolactone treatment on serum low-density lipoprotein cholesterol. The concentrations of serum low-density lipoprotein cholesterol (mmol/L) are measured before and after spironolactone treatment, respectively. The changes of serum low-density lipoprotein cholesterol are analyzed after the spironolactone treatment.
Change of serum creatinine | From enrollment to spironolactone treatment at 12 months.
  This study will gain insight into the effect of spironolactone treatment on serum creatinine. The concentrations of serum creatinine (µmol/L) are measured before and after spironolactone treatment, respectively. The changes of serum creatinine are analyzed after the spironolactone treatment.
Change of 24-hour urine microalbumin | From enrollment to spironolactone treatment at 12 months.
  This study will gain insight into the effect of spironolactone treatment on 24-hour urine microalbumin. The concentrations of 24-hour urine microalbumin (mg) are measured before and after spironolactone treatment, respectively. The changes of 24-hour urine microalbumin are analyzed after the spironolactone treatment.
Change of estimated glomerular filtration rate | From enrollment to spironolactone treatment at 12 months.
  This study will gain insight into the effect of spironolactone treatment on estimated glomerular filtration rate. The variables of estimated glomerular filtration rate (ml/min/1.73m²) are measured before and after spironolactone treatment, respectively. The changes of estimated glomerular filtration rate are analyzed after the spironolactone treatment.
Change of urine albumin-to-creatinine ratio | From enrollment to spironolactone treatment at 12 months.
  This study will gain insight into the effect of spironolactone treatment on urine albumin-to-creatinine ratio. The variables of urine albumin-to-creatinine ratio (mg/g) are measured before and after spironolactone treatment, respectively. The changes of urine albumin-to-creatinine ratio are analyzed after the spironolactone treatment.
Change of urine aldosterone | From enrollment to spironolactone treatment at 12 months.
  This study will gain insight into the effect of spironolactone treatment on urine aldosterone. The concentrations of urine aldosterone (ng/dL) are measured before and after spironolactone treatment, respectively. The changes of urine aldosterone are analyzed after the spironolactone treatment.
Incidence of cardiovascular events | From enrollment to spironolactone treatment at 12 months.
  This study will gain insight into the effect of spironolactone treatment on cardiovascular events (%). The cardiovascular events include coronary heart disease, stroke, peripheral artery disease, etc. Incidence of cardiovascular events are analyzed after the spironolactone treatment.
Numbers of adverse reactions | From enrollment to spironolactone treatment at 12 months.
  This study will evaluate the adverse effects of spironolactone treatment. The adverse reactions include itchy skin, tiredness, headache, etc. Numbers of adverse reactions are analyzed after the spironolactone treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Zhu, MD, Study Chair — Department of Hypertension and Endocrinology, Daping Hospital, Army Medical University
Locations (1):
- Daping Hospital, Army Medical Center of PLA, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No